CLINICAL TRIAL: NCT00002535
Title: TUMOR INFILTRATING LYMPHOCYTE THERAPY FOR ADVANCED MELANOMA USING IMMUNOMODULATION, A PHASE II STUDY
Brief Title: Indomethacin Plus Biological Therapy in Treating Patients With Advanced Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Luke's Medical Center (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: STLMC-BRM-93004; CDR0000078467 (Registry Identifier: PDQ (Physician Data Query)); NCI-V93-0295
Record Dates: First submitted 1999-11-01; First posted 2004-07-29 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2000-08

CONDITIONS: Melanoma (Skin)
Keywords: stage III melanoma; stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — aldesleukin; Cyclophosphamide; Indomethacin

INTERVENTIONS:
Biological: aldesleukin
Biological: lymphokine-activated killer cells
Biological: therapeutic tumor infiltrating lymphocytes
Drug: cyclophosphamide
Drug: indomethacin

SUMMARY:
RATIONALE: Biological therapies use different ways to stimulate the immune system and stop tumor cells from growing. Combining biological therapies with indomethacin and cyclophosphamide may kill more tumor cells.

PURPOSE: Phase II trial to compare the effectiveness of indomethacin and biological therapy with or without cyclophosphamide in treating patients who have advanced melanoma that has not responded to previous therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine whether indomethacin given prior to tumor removal can increase the number of tumor infiltrating lymphocytes (TIL) obtained from the tumor specimen of patients with advanced melanoma. II. Determine the efficacy of administering concurrent indomethacin to maximize immune effector cell function in situ during interleukin-2/TIL therapy in these patients. III. Determine the relationship between the phenotypic character of TIL (generated in culture from the patient's tumor) and the response to therapy. IV. Correlate the lytic activity or lymphokine production of TIL (generated in culture from the patient's tumor) with clinical response to therapy. V. Generate and use lymphokine-activated killer (LAK) cells in those patients who do not have TIL available for therapy and evaluate LAK cells in the same manner as TIL.

OUTLINE: Patients with resectable tumors and with adequate generation of TIL are treated on Regimen A; those with unresectable tumors or insufficient TIL are treated on Regimen B. The following acronyms are used: CTX Cyclophosphamide, NSC-26271 IL-2 Interleukin-2 (Cetus), NSC-373364 LAK Lymphokine-Activated Killer Cells TIL Tumor Infiltrating Lymphocytes Regimen A: Prostaglandin Inhibition Therapy plus Biological Response Modifier Therapy. Indomethacin; plus CTX; IL-2-activated TIL; IL-2. Regimen B: Prostaglandin Inhibition Therapy plus Biological Response Modifier Therapy. Indomethacin; plus IL-2-activated LAK; IL-2.

PROJECTED ACCRUAL: Up to 30 patients will be accrued over 3 years. If 0 of the first 10 patients, no more than 1 of the first 15 patients, or no more than 2 of the first 20 patients respond, accrual will cease.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically documented melanoma that is metastatic or unresectable and unresponsive to conventional chemotherapy and/or radiotherapy Measurable or evaluable disease required Measurable disease defined as bidimensionally measurable lesion on physical exam, x-ray, or MRI Evaluable disease defined as: Unidimensionally measurable lesion on x-ray, scan, or photograph Disease assessable by serial chemistries, tumor markers, or nonspecific scans Disease assessable by functional manifestations (e.g., change in performance status, 10% or greater change in weight) Previously irradiated lesion with subsequent disease progression documented Bone-only lesions may be considered evaluable (lytic lesion on x-ray or bone scan should be followed) No metastases on CT or MRI involving more than 50% of the liver No uncontrolled or untreated CNS metastases

PATIENT CHARACTERISTICS: Age: Over 16 Performance status: ECOG 0 or 1 Life expectancy: At least 3 months Hematopoietic: (unless tumor involvement of bone marrow or spleen is documented) WBC at least 3,500/mm3 Absolute granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 11.5 g/dL No significant hematologic abnormalities Hepatic: (unless tumor involvement of liver is documented) Bilirubin no greater than 1.6 mg/dL SGOT no greater than 150 U/L PT at least 1.5 times control PTT less than 1.5 times control Renal: (unless tumor involvement of kidney is documented) Creatinine no greater than 2.0 mg/dL Creatinine clearance at least 50 mL/min Calcium no greater than 12 mg/dL No symptomatic hypercalcemia Cardiovascular: No myocardial infarction within 6 months No congestive heart failure No edema No hypotension or hypertension No coronary artery disease No history of arrhythmia No contraindication to the use of pressor agents Pulmonary: FEV1 at least 65% of predicted Other: No significant organ dysfunction No uncontrolled bacterial, viral, or fungal infection No active peptic or duodenal ulcer No psychiatric or seizure disorder No prior solid organ allograft HIV and hepatitis B surface antigen seronegative within 6 months of study entry No second malignancy within 5 years except: Inactive nonmelanomatous skin cancer Carcinoma in situ of the cervix No other serious illness that would limit survival to less than 2 years Negative pregnancy test

PRIOR CONCURRENT THERAPY: Biologic therapy: More than 4 weeks since immunotherapy Chemotherapy: Prior anthracyclines allowed provided no symptomatic heart disease is present More than 4 weeks since chemotherapy (at least 2 weeks, with recovery, if disease progression is documented) More than 6 weeks since nitrosoureas, melphalan, or mitomycin Endocrine therapy: More than 1 week since corticosteroids (except physiological doses for respiratory ailments or adrenal insufficiency) Radiotherapy: More than 4 weeks since radiotherapy (at least 2 weeks, with recovery, if disease progression is documented) Surgery: More than 3 weeks since major surgery (excluding surgery for tumor collection)

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1993-07; Study Completion 2004-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John P. Hanson, MD, Study Chair — St. Luke's Medical Center
Locations (1):
- St. Luke's Medical Center, Milwaukee, Wisconsin, United States